CLINICAL TRIAL: NCT06361368
Title: Efficacy Assessment of Probiotics in Improving Sleep Indices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYCU112174AF
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-03

CONDITIONS: Insomnia
Keywords: PS150; Probiotics; Circadian Rhythm; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS150 (Experimental): Each PS150 (Limosilactobacillus fermentum) capsule contained 5 × 10^9 colony forming units (CFU) , 1 capsule daily use.
  Interventions: Dietary Supplement: PS150
- Placebo (Placebo Comparator): The placebo capsule contains microcrystalline cellulose, 1 capsule daily use.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PS150 — Participants took one capsule with PS150 after dinner for 30 days.
  Other Names: Limosilactobacillus fermentum
  Arms: PS150
Dietary Supplement: Placebo — Participants took one capsule with placebo after dinner for 30 days.
  Arms: Placebo

SUMMARY:
To determine whether PS150 (1) reduces insomnia symptoms, (2) improves sleep quality, (3) adjusts autonomic nervous system functioning, (4) reduces the severity of anxiety and depressive symptoms, and (5) adjusts microbiome and endocrine functions.

DETAILED DESCRIPTION:
One-hundred-forty participants with self-reported insomnia (PSQI≥ 7 & 22 > ISI ≥ 12) aged between 20 and 60 years old are estimated to be recruited and randomly assigned to two arms, the PS150 group and the placebo group, under the double-blinded trial. Participants take one capsule of probiotics or placebo after dinner for 30 days. Study measures include polysomnography (PSG), subjective sleep, depressive, and anxiety questionnaires, sleep diary, fecal sampling, saliva testing, and urine testing.

ELIGIBILITY:
Inclusion Criteria:

1. aged 20-60 years old,
2. self-reported Insomnia (PSQI ≥ 7 & 22 > ISI ≥ 12),
3. 17.5 < BMI < 35 kg/m^2, and
4. regular sleep cycle.

Exclusion Criteria:

1. used antibiotic, sleep aids, tranquilizers, or antipsychotic treatment within the last month,
2. used other probiotic products within the last month,
3. taking medications known to commonly induce sleep disorders (such as corticosteroids, antihistamines, and stimulants, etc.) or currently undergoing hormone therapy, including contraceptive pills,
4. have undergone hepatobiliary gastrointestinal tract surgery
5. lactic acid bacteria allergy,
6. with cancer, cardiovascular disease, psychiatric illness, or kidney disease,
7. with uncontrolled diabetes mellitus or hypertension,
8. with sleep disorders other than insomnia,
9. allergic to lactobacillus,
10. reported tobacco, alcohol, caffeine or drug addiction,
11. traveled to different time zone in long-distance trip within the last month,
12. participated in other interventional studies within the last three months, and
13. evaluated as unsuitable participant by PI.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (PSG) | Baseline, day30
  According to the polysomnography, we can analysis participants' brain waves (alpha,beta,theta,delta), sleep stages, and autonomic nervous system functioning to evaluate their objective sleep quality.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline, day 30
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated inventory that assesses sleep quality over the past 1-month. The measure consists of 19 individual items, creating 7 components that produce one global score. It takes 5-10 minutes to complete.The maximum global score is 21. A higher score reflects more poor sleep quality.
Insomnia Severity Index (ISI) | Baseline, day 30
  The Insomnia Severity Index (ISI) is designed as a brief screening tool for insomnia. The seven-item questionnaire asks respondents to rate the nature and symptoms of their sleep problems using a 5-Likert scale. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia.The maximum total score is 28.
Beck Depression Inventory-Second Edition (BDI-II) | Baseline, day 30
  The Beck Depression Inventory-Second Edition (BDI-II) is a 21-item, self-rated inventory that evaluates key symptoms of depression. It rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. A higher score reflects greater symptoms of depression.
Beck Anxiety Inventory (BAI) | Baseline, day 30
  The Beck Anxiety Inventory (BAI) is a 21-item, self-rated inventory that evaluates anxiety levels. It rated on a scale from 0 to 3. Each item is descriptive of subjective, somatic, or panic-related anxious symptoms.The maximum total score is 63. A higher score reflects greater symptoms of anxiety.
VAS-Sleep | Baseline, day 30
  Visual Analogue Scale (VAS) consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).
Epworth Sleepiness Scale (ESS) | Baseline, day 30
  The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of sleepiness. It is a list of eight situations in which you rate your tendency to become sleepy. Each item is rated on the scale from 0, no chance of dozing, to 3, high chance of dozing.
Stanford Sleepiness Scale (SSS) | Baseline, day 30
  The Stanford Sleepiness Scale (SSS) is a 7-point Likert inventory to evaluate a respondent's sleepiness at the time when it is completed.
Visual Analogue Scale for gastrointestinal symptoms (VAS-GI) | Baseline, day 30
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in respondents before and after taking PS150 or Placebo.
Saliva Melatonin | Baseline, day 30
  pg/ml of melatonin in saliva measured by enzyme-linked immunosorbent assay.
Saliva Cortisol | Baseline, day 30
  Cortisol is a steroid hormone that is produced by the adrenal glands which sit on top of each kidney. When released into the bloodstream, cortisol can act on many different parts of the body and can help:
  body respond to stress or danger increase your body's metabolism of glucose control your blood pressure reduce inflammation. Cortisol is also needed for the fight or flight response which is a healthy, natural response to perceived threats. The amount of cortisol produced is highly regulated by your body to ensure the balance is correct.
Saliva Interleukin-6 (IL-6) | Baseline, day 30
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80°C. Enzyme-linked immunosorbent assays were used to quantify IL-6 amount (ng/mL).
Saliva Total Antioxidant Capacity (TAC) | Baseline, day 30
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80°C. Enzyme-linked immunosorbent assays were used to quantify TAC amount (nmol/mL).
Saliva Serotonin | Baseline, day 30
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80°C. Enzyme-linked immunosorbent assays were used to quantify serotonin amount (ng/mL).
Saliva gamma-aminobutyric acid (GABA) | Baseline, day 30
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80°C. Enzyme-linked immunosorbent assays were used to quantify GABA amount (pg/mL).
Saliva Orexin | Baseline, day 30
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80°C. Enzyme-linked immunosorbent assays were used to quantify Orexin amount.
Urine 6-sulfatoxymelatonin | Baseline, day 30
  In order to determine the levels of 6-sulphatoxymelatonin from patients in the experimental and control groups, urine samples will be taken between between 21:00 to 23:00 at night. A urine sample will be taken into a sample container containing 10-15 ml of 6 M hydrochloric acid (HCl) and stored at -80 degrees for analysis in the biochemistry laboratory.
Urine Norepinephrine | Baseline, day 30
  In order to determine the levels of norepinephrine from patients in the experimental and control groups, urine samples will be taken between between 21:00 to 23:00 at night. A urine sample will be taken into a sample container containing 10-15 ml of 6 M hydrochloric acid (HCl) and stored at -80 degrees for analysis in the biochemistry laboratory.
Actigraphy | Baseline, day 30
  Actigraph will be placed on the non-dominant wrist and activities will be monitored continuously and recorded at one minute intervals during wakefulness and sleep.
  The times of wakefulness and sleep will be determined individually through a diary kept by the participants, together with the times calculated by the actigraph monitor.
  The participants will keep the device for a period of 7 days before and the last 7-day of training session. The device will be removed only at bath time and replaced to the wrist immediately after.
Sleep Diary | Baseline, day 30
  The sleep diary is a daily self-reported 12-item form within 30 minutes after wake up. It assesses respondent's time taken to fall asleep (sleep onset latency), wake after sleep onset, total sleep, total time in bed, and sleep efficiency, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl C Yang, doctor, Study Chair — Institute of Brain Science ,National Yang Ming Chiao Tung University, Taipei City, Taiwan
Locations (1):
- Institute of Brain Science National Yang Ming Chiao Tung University, Taipei, Taiwan